CLINICAL TRIAL: NCT06986473
Title: Innovating a Questionnaire to Investigate the Awareness of Dermatologists Regarding the Role of Physical Therapy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ola galal eldemerdash sakr, Demonestrator, Cairo University
Other Study IDs: P.T.REC/012/005402
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-10

CONDITIONS: Measure the Level of Awareness of Dermatologists
Keywords: physical therapy; dermatologists; skin diseases; referral practices; interprofessional collaboration; awareness; Egypt; Questionnaire
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

INTERVENTIONS:
Other: Questionnaire that measure the level of awareness of dermatologists — This study will be an observational cross-sectional analytical study that will recruit 165 dermatologists of both genders according to sample size calculation from different outpatient clinics in Cairo teaching hospitals. The aim of the study will be to develope a questionnaire to evaluate the awareness of Egyptian dermatologist towards the role of physical therapy in patients with various skin diseases

SUMMARY:
The purpose of this study will be developing a questionnaire to evaluate the level of awareness of dermatologists regarding the role of physical therapy in patients with different skin diseases.

BACKGROUND:

Skin diseases encompass a wide range of conditions that affect the skin, hair, and nails. They can be acute or chronic, benign or malignant, and can significantly impact an individual's quality of life. Understanding the epidemiology, causes, types, prevalence, and treatment options of skin diseases is crucial for effective management and improving patient outcomes, especially in regions like the Middle East and Egypt.

The treatment of skin diseases in the Middle East and Egypt involves a combination of topical and systemic therapies, lifestyle modifications, and sometimes surgical interventions. While treatments can be effective, they may also have side effects

Physical therapy plays a significant and often underappreciated role in the management of various skin diseases. While traditionally associated with musculoskeletal and neurological conditions, it can also be beneficial in treating and managing skin-related disorders

ELIGIBILITY:
Inclusion Criteria:

* Dermatologists that will be included in the study will be with;

  1. Professional Status: Must be a certified dermatologist.
  2. Location: Must be practicing in Cairo teaching hospitals.
  3. Active Practice: Must currently be practicing either in a clinical setting, hospital, or private practice.
  4. Consent: Must provide informed consent to participate in the study.
  5. Experience: Dermatologists of more than 5 years of experience.

     Exclusion Criteria:
* This study will exclude dermatologists with the following criteria;

  1. Non-Dermatologists: Professionals who are not dermatologists, such as general practitioners, nurses, or other healthcare providers who do not specialize in dermatology.
  2. Inactive Professionals: Dermatologists who are retired or currently not practicing for any reason (e.g., on extended leave).
  3. Non-Consenting Individuals: Individuals who do not agree to participate in the study or who do not provide informed consent.
  4. Incomplete Surveys: Participants who do not complete the entire survey or interview process, depending on the data collection method used in the study.
  5. Non-Egyptian Practitioners: Dermatologists practicing outside of Egypt, even if they are Egyptian nationals, to maintain a focus on the practices and awareness within the Egyptian healthcare system

Min Age: 24 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Dermatologists from Cairo teaching hospitals
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Level of awareness of Egyptian dermatologists | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy Cairo university in Egypt, Giza, Egypt